CLINICAL TRIAL: NCT04008732
Title: A Single Centre, Open-label, Randomised, Single Dose, Six Period, Reference Replicate, Crossover Study to Evaluate the Bioavailability of MED2005
Brief Title: Evaluating MED2005 & Nitrostat Bioavailability
Acronym: FM58
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Futura Medical Developments Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: FM58
Record Dates: First submitted 2018-01-24; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Nitroglycerin; Administration, Sublingual

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- MED2005 (0.6 mg) (Experimental): MED2005 (0.2% GTN) gel to be used topically in Part 1 of the study
  Interventions: Drug: MED2005; Drug: Nitrostat 0.6Mg Sublingual Tablet
- MED2005 (1.2 mg) (Experimental): MED2005 (0.4% GTN) gel to be used topically in Part 1 of the study
  Interventions: Drug: MED2005; Drug: Nitrostat 0.6Mg Sublingual Tablet
- MED2005 (1.8 mg) (Experimental): MED2005 (0.6% GTN) gel to be used topically in Part 1 of the study
  Interventions: Drug: MED2005; Drug: Nitrostat 0.6Mg Sublingual Tablet
- Nitrostat (1.8 mg) - Treatment Period 1 (Active Comparator): 3 x 0.6 mg tablets will be required to make up the 1.8 mg dose to be used orally in Part 1 of the study but to be dosed in two treatment periods
  Interventions: Drug: MED2005; Drug: Nitrostat 0.6Mg Sublingual Tablet
- Nitrostat (1.8 mg) - Treatment Period 2 (Active Comparator): 3 x 0.6 mg tablets will be required to make up the 1.8 mg dose to be used orally in Part 1 of the study but to be dosed in two treatment periods
  Interventions: Drug: MED2005; Drug: Nitrostat 0.6Mg Sublingual Tablet
- MED2005 (2.4 mg)- Part 1 (Experimental): MED2005 (0.8% GTN) gel to be used topically in Part 1 of the study
  Interventions: Drug: MED2005; Drug: Nitrostat 0.6Mg Sublingual Tablet
- Intravenous (I.V.) dose of GTN (0.3 mg) (Active Comparator): GTN solution for infusion (1 mg/ml) to be used intravenously in Part 2 of the study
  Interventions: Drug: Nitro Pohl
- MED2005 (2.4 mg)- Part 2 (Experimental): MED2005 (0.8% GTN) gel to be used topically in Part 2 of the study
  Interventions: Drug: Nitro Pohl

INTERVENTIONS:
Drug: MED2005 — (Day -1 to Day 1): Subjects will undergo six treatment periods, each separated by at least a two day washout. Each treatment period will be approximately 1 day in duration from the afternoon of Day -1 to the afternoon of Day 1 at 6 hours (h) post-dose. In each of the treatment periods, the subject will receive one of the six administrations over 6 treatment periods (1/period) and will return approximately two days later for the next treatment period.
  Other Names: glyceryl trinitrate
  Arms: MED2005 (0.6 mg); MED2005 (1.2 mg); MED2005 (1.8 mg); MED2005 (2.4 mg)- Part 1; Nitrostat (1.8 mg) - Treatment Period 1; Nitrostat (1.8 mg) - Treatment Period 2
Drug: Nitrostat 0.6Mg Sublingual Tablet — Active comparator to be used for Part 1 of the study. Nitrostat will be dosed in two treatment periods and 3 x 0.6 mg tablets will be required to make up the 1.8 mg dose.
  Other Names: Nitroglycerin 0.6 mg
  Arms: MED2005 (0.6 mg); MED2005 (1.2 mg); MED2005 (1.8 mg); MED2005 (2.4 mg)- Part 1; Nitrostat (1.8 mg) - Treatment Period 1; Nitrostat (1.8 mg) - Treatment Period 2
Drug: Nitro Pohl — to be dosed intravenously in Part 2 of the study
  Other Names: Nitroglycerin
  Arms: Intravenous (I.V.) dose of GTN (0.3 mg); MED2005 (2.4 mg)- Part 2

SUMMARY:
Futura Medical Developments Ltd (FMD) are developing a gel formulation of GTN (MED2005) as a topical treatment for ED delivered using DermaSys®, a versatile and bespoke technology. Treatment requires the application of a small quantity of gel (approx 300 mg), containing a fixed dose of GTN, to the glans of the penis. Pharmacokinetic studies in healthy volunteers indicate rapid absorption of the drug and low systemic exposure, reducing the risk of adverse events (such as headache) commonly associated with GTN therapy.

The purpose of this study is to demonstrate similar or lower bioavailability of GTN from MED2005 (test IMP) with that from Nitrostat (reference IMP).

The study will be conducted in two parts (Part 1 and 2). Part 1 will be conducted in 30 subjects and Part 2 will be conducted in 10 subjects. Part 1 will compose of a pre-study screen, followed by six treatment periods and a post-study follow-up.

Part 2 will compose of a pre-study screen, followed by two treatment periods and a post-study follow-up. Subjects can only participate in either Part 1 or 2 of the study (not both).

DETAILED DESCRIPTION:
GTN is a well-established vasodilatory therapeutic agent with a long, documented history of use and comprehensive safety profile. In Europe, licensed indications for GTN include the treatment and prophylaxis of angina pectoris and the relief of pain associated with chronic anal fissure. Other indications for prescription only parenteral products include use during cardiac surgery and for emergency reduction of blood pressure.

GTN's vasodilatory action is thought to result from the release of nitric oxide (NO) in vascular smooth muscle. NO stimulates guanylate cyclase, the enzyme responsible for production of cGMP, whose action is to lower intracellular calcium resulting in smooth muscle relaxation and vasodilation.

In the case of erectile dysfunction, GTN works locally by penetrating the glans/penile skin and directly targeting penile blood vessels. Nitrates appear to have a direct, local effect on penile haemodynamics. The most likely mechanism for the erectile effect of nitrates involves nitrate induced dilation of the cavernous and helicine arteries, thereby increasing blood flow to the lacunar spaces, coupled with nitrate-induced relaxation of trabecular smooth muscle.

Nitroglycerin (Nitrostat) is indicated for the acute relief of an attack or acute prophylaxis of angina pectoris due to coronary artery disease.

The principal pharmacological action of nitroglycerin is relaxation of vascular smooth muscle. Although venous effects predominate, nitroglycerin produces, in a dose-related manner, dilation of both arterial and venous beds. Dilation of postcapillary vessels, including large veins, promotes peripheral pooling of blood, decreases venous return to the heart, and reduces left ventricular end-diastolic pressure (preload). Nitroglycerin also produces arteriolar relaxation, thereby reducing peripheral vascular resistance and arterial pressure (afterload), and dilates large epicardial coronary arteries; however, the extent to which this latter effect contributes to the relief of exertional angina is unclear.

Nitroglycerin forms free radical nitric oxide (NO) which activates guanylate cyclase, resulting in an increase of guanosine 3'5' monophosphate (cyclic GMP) in smooth muscle and other tissues. These events lead to dephosphorylation of myosin light chains, which regulate the contractile state in smooth muscle, and result in vasodilatation.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between 18 and 50 years of age, inclusive (at screening).
2. A BMI of 18.5-30 kg/m2 (inclusive).
3. No clinical significant abnormal serum biochemistry, haematology and urine examination values as defined by the Investigator.
4. A negative urinary drugs of abuse screen. A positive alcohol test may be repeated on admission at the discretion of the Investigator.
5. Negative HIV and Hepatitis B and C results.
6. No clinically significant abnormalities in 12-lead ECG as defined by the Investigator.
7. No clinically significant deviation outside the normal ranges for blood pressure and heart rate measurements as defined by the Investigator (please refer to appendix 1 for normal ranges).
8. Subjects (unless anatomically sterile (documented evidence) or where abstaining from sexual intercourse is in line with the preferred and usual lifestyle of the subject) and sexual partners must use 2 effective contraception methods during the trial and for 3 months after the last dose, for example:

   * Oral contraceptive + condom.
   * Intra-uterine device (IUD) + condom.
   * Diaphragm with spermicide + condom.
9. Subjects must be available to complete all periods of the study and the follow-up visit.
10. Subjects must satisfy the PI / designee about their fitness to participate in the study.
11. Subjects must be able to read and understand the informed consent form and must provide written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant history of gastrointestinal disorder likely to influence IMP absorption (Part 1 only).
2. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 28 days (or 5 half-lives (whichever is longer) prior to the first dose of IMP, unless in the opinion of the Investigator and Sponsor's Responsible Physician the medication will not interfere with the study procedures or compose subject safety.
3. Evidence of renal, hepatic, central nervous system, respiratory, cardiovascular or metabolic dysfunction.
4. A clinically significant history of drug or alcohol abuse within 2 years before the first dose of IMP.
5. A clinically significant history of previous allergy/sensitivity to GTN, other nitrates and/or any of the excipients in either the test of reference products.
6. Recent history of using PDE5 inhibitors or alkyl nitrates (e.g. poppers).
7. A history of frequent tension headaches or vascular headaches or migraine.
8. A history of increased intra-cranial pressure or spinal cord injury.
9. A history of severe psychological disorders.
10. A presence of scarring/piercings/tattoos at the site of MED2005 administration (penis) (or any other features that the Investigator considers may influence IMP absorption).
11. Subjects (if uncircumcised) who are not able to retract foreskin of penis easily without any discomfort.
12. Any obvious sensitivity/local tolerability issues at the site of medication application.
13. Inability to communicate well with the investigator (i.e. language problems, poor mental development or impaired cerebral function).
14. Participation in a New Chemical Entity or marketed drug clinical study within the previous 3 months or, five half-lives of study drug, whichever is the longer period. (NB. the three month washout period between trials is defined as the period of time elapsed between the last dose of the previous study and the first dose of the next study).
15. Subjects who smoke (or ex-smokers) who have smoked or used nicotine-containing products (including snuff, chewing tobacco, cigars, pipes or nicotine replacement products) within four months prior to first dose.
16. Donation or receipt of ≥ 450 mL of blood within 3 months before the first dose of IMP.
17. Donation of sperm from the first dose and for at least 3 months after the last dose of IMP.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Yes
Enrollment: 40 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
To demonstrate similar or lower bioavailability of GTN when administered as a gel via MED2005 compared to Nitrostat (which will administrated as a sublingual tablet) in terms of AUC0-t (Part 1) | 22 days
  The primary objective of this human pharmacology study is to demonstrate similar or lower bioavailability of GTN
To demonstrate similar or lower bioavailability of GTN when administered as a gel via MED2005 compared to Nitrostat (which will administrated as a sublingual tablet) in terms of AUC0-inf (Part1) | 22 days
  The primary objective of this human pharmacology study is to demonstrate similar or lower bioavailability of GTN
To demonstrate similar or lower bioavailability of GTN when administered as a gel via MED2005 compared to Nitrostat (which will administrated as a sublingual tablet) in terms of Cmax (part1) | 22 days
  The primary objective of this human pharmacology study is to demonstrate similar or lower bioavailability of GTN

SECONDARY OUTCOMES:
The pharmacokinetics of GTN metabolite 1,2-GDN will be evaluated following the administration of MED2005 compared with Nitrostat (Part 1). | 22 days
  The percentage of drug metabolites in the bloodstream following administration of MED2005 (test formulation) with Nitrostat (reference) (part 1) will be compared and evaluated.
Adverse events (AEs) coded using Medical Dictionary for Regulatory Activities (MedDRA) version 20.0 or higher | 46 days
  The incidence of treatment-emergent AEs (TEAE) will be summarised by organ system, preferred term, severity and relationship to study drug. AEs will be identified via abnormal vital signs, abnormal 12-lead ECG parameters, and/or abnormal laboratory safety data
GTN absorption (to quantify the amount of GTN remaining on the glans penis post application) | 10 days
  To quantify the amount of GTN remaining on the glans penis post application of MED2005 (Part 2).
GTN absorption (to quantify a figure of 100% GTN being absorbed) | 10 days
  I.V. dosing to quantify a figure of 100% GTN being absorbed (Part 2).
The pharmacokinetics of GTN metabolite1,3-GDN will be evaluated following the administration of MED2005 compared with Nitrostat (Part 1). | 22 days
  the percentage of drug metabolites in the bloodstream following administration of MED2005 (test formulation) with Nitrostat (reference) (part 1) will be compared and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Israel, Israel, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, Wales, United Kingdom

IPD SHARING:
Plan to Share IPD: No